CLINICAL TRIAL: NCT05262907
Title: Assessment of Ventricular Volumes and Function in Single Ventricle Patients Using Ventripoint 3D Echocardiography
Brief Title: Ventripoint Single Ventricle Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00108548
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Congenital Heart Disease; Single-ventricle
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Ventripoint 3D Echocardiogram (Experimental): Ventripoint 3D Echo performed on subject to validate technology for use in single ventricle patients.
  Interventions: Device: Ventripoint Echocardiogram
- Transthoracic Echocardiogram or Cardiac MRI (Active Comparator): Non-invasive imaging of the heart to evaluate structure and function.
  Interventions: Device: Transthoracic Echocardiogram or Cardiac MRI

INTERVENTIONS:
Device: Transthoracic Echocardiogram or Cardiac MRI — Non-invasive imaging of the heart to evaluate structure and function.
  Arms: Transthoracic Echocardiogram or Cardiac MRI
Device: Ventripoint Echocardiogram — Non-invasive ultrasound of the heart to evaluate structure and function through 3D imaging.
  Arms: Ventripoint 3D Echocardiogram

SUMMARY:
This study will validate a coordinate-based 3-dimensional echocardiographic technique for the assessment of cardiac size and function in children and young adults with functional single ventricles.

DETAILED DESCRIPTION:
The accuracy of current echocardiographic techniques for measuring ventricular size and function are limited by geometric assumptions, which are particularly problematic in malformed hearts or functional single ventricles, as well as the inability to visualize the entire heart at one time from a single imaging window, and higher heart rates degrading 3D imaging volume rates. This study will validate a coordinate-based 3-dimensional echocardiographic technique for the assessment of cardiac size and function in children and young adults with functional single ventricles, including a comparison to the gold standard of cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

* All patients with functional single ventricles will be included, regardless of age or surgical palliation stage, who have had or are having a clinically ordered transthoracic echocardiogram and/or cardiac MRI.

Exclusion Criteria:

* Patients with congenital heart disease other than functional single ventricles, patients with single ventricle physiology (but not single ventricle anatomy) following a biventricular conversion pathway, or patients unable to understand or consent in English will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Cardiac function of the right ventricle as measured by ejection fraction | Day 1
  Ejection Fraction (EF) is a measurement of the percentage of blood leaving your heart each time it squeezes (contracts)with each heart beat.
Cardiac function of the left ventricle as measured by ejection fraction | Day 1
  Ejection Fraction (EF) is a measurement of the percentage of blood leaving your heart each time it squeezes (contracts)with each heart beat.
Right ventricular dimension as measured by end diastolic volume | Day 1
  End Diastolic Volume (EDV) is the volume of blood in a ventricle at end load or filling in (diastole) or the amount of blood in the ventricles just before systole.
Right ventricular dimension as measured by end systolic volume | Day 1
  End Systolic Volume (ESV) is the volume of blood in a ventricle at the end of contraction, or systole, and the beginning of filling, or diastole.
Left Ventricular Dimension as measured by end diastolic volume | Day 1
  End Diastolic Volume (EDV) is the volume of blood in a ventricle at end load or filling in (diastole) or the amount of blood in the ventricles just before systole.
Left Ventricular Dimension as measured by end systolic volume | Day 1
  End Systolic Volume (ESV) is the volume of blood in a ventricle at the end of contraction, or systole, and the beginning of filling, or diastole.
Left Ventricular Dimension as measured by end diastolic diameter | Day 1
  End Diastolic Diameter (EDD) is the diameter across the left ventricle of the heart at the end of diastole, that is, when the heart muscle is maximally relaxed, and usually corresponds to its largest diameter.
Left Ventricular Dimension as measured by end systolic diameter | Day 1
  End Systolic Diameter (ESD) is the diameter across the left ventricle of the heart at the end of systole, that is, when the heart muscle is maximally contracted, and usually corresponds to its smallest diameter.
Right Ventricular Function as measured by tricuspid annular plane systolic excursion | Day 1
  Tricuspid Annular Plane Systolic Excursion (TAPSE) is a measurement of the decent of the right ventricular base towards a relatively fixed apex.
Right Ventricular Function as measured by myocardial performance index | Day 1
  RV Myocardial Performance Index (MPI) is a measurement that incorporates tricuspid valve closure to opening time and right ventricular ejection time to evaluate efficiency of the ventricle.
Left Ventricular Function as measured by myocardial performance index | Day 1
  LV Myocardial Performance Index (MPI) is a measurement that incorporates mitral valve closure to opening time and left ventricular ejection time to evaluate efficiency of the ventricle.
Left Ventricular Function as measured by tissue doppler imaging | Day 1
  Tissue Doppler Imaging (TDI) a measurement of the velocity of myocardial motion.
Left ventricular function as measured by shortening fraction | Day 1
  Shortening fraction(SF) is a measurement of the percentage of change in left ventricular diameter during systole.
Presence of ventricular dysfunction as measured by strain | Day 1
  Strain is a measure of deformity in the muscle of the ventricle.

CONTACTS AND LOCATIONS:
Overall Officials: Piers Barker, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No